CLINICAL TRIAL: NCT06365138
Title: Analysis of Individual Activity at the Time of Aortic Rupture in Patients With Abdominal Aortic Aneurysms
Status: Recruiting | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Collaborators: Epidemiology, Medical Faculty, University Augsburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: Aortic Rupture
Record Dates: First submitted 2024-01-29; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Aortic Aneurysm
Keywords: Aortic Rupture; Physical stress; Emotional Stress; Rupture Risc; Follow-Up; Activity
MeSH Terms: conditions — Aortic Aneurysm; Aortic Rupture; Stress, Psychological; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Bahaviour at the time of an aortic aneurysm rupture — Questionnaire and patient interview, diary for day of rupture and the three previous days

SUMMARY:
It is currently unclear what activities aneurysms are involved in at the time of rupture. The aim of the study is to determine the activity performed at the time of aneurysm rupture.

DETAILED DESCRIPTION:
The scientifically proven risk factors that significantly favor the rupture of an aortic aneurysm are female gender, the maximum diameter of the aortic aneurysm and the patient's current smoking status.

However, no analysis of the occupation performed at the time of aortic rupture of an abdominal aortic aneurysm has yet been carried out.

High arterial systolic blood pressure can promote aortic rupture. Blood pressure peaks can occur during physical exertion, for example when lifting heavy loads or during defecation.

Patients with an existing intact aortic aneurysm are currently advised to avoid such behaviors as a preventive measure. This includes, among other things, the practice of strength training or certain types of sport. This can subsequently lead to a reduction in quality of life, although this cannot currently be substantiated by scientific data. There is also no current guideline recommendation in this regard.

Furthermore, the role of stress and / or emotionally stressful events in connection with the occurrence of aortic ruptures has not yet been recorded in the literature. There is work on this in connection with aortic dissections, which postulates that an increase in emotional or psychological stress can lead to acute hypertension, which can cause a previously damaged aorta to rupture. A similar pathomechanism would also be conceivable for the rupture of aortic aneurysms.

There are indications that, in addition to gender-specific differences in the occurrence of aortic ruptures, there is also a different risk of rupture based on certain pre-existing conditions, dietary habits and age.

ELIGIBILITY:
Inclusion Criteria:

* inclusion of all patients with ruptured aortic aneurysm in Augsburg University Hospital
* Written consent to participate in the study by the patient or their legal representative

Exclusion Criteria:

* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ruptured aortic aneurysm in Augsburg University Hospital form 01/01/24 till 12/31/29 for the prospecitve part of the trial.
  All patients who have been treated for a ruptured aortic aneurysm in Augsburg University Hospital form 01/01/13 till 12/31/23 for the retrospectitve part of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Occupation at the time of the aortic aneurysm rupture | Occupation at the day of the aortic rupture and the three days prior
  Occupation at the time of the aortic aneurysm rupture

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Duerr, Prof., Study Chair — University Hospital Augsburg Vascular Surgery
Locations (1):
- University Hospital Augsburg, Augsburg, Germany